CLINICAL TRIAL: NCT06647043
Title: A Single-arm, Open-label Clinical Trial to Evaluate the Effect of SMT04 Pro in Irritable Bowel Syndrome (IBS)
Brief Title: Evaluate the Effect of Synbiotics in Irritable Bowel Syndrome
Acronym: IBSXtra02
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Collaborators: GenieBiome Limited (Industry)
Responsible Party: Principal Investigator, Lee Yeong Yeh, Professor Dr, Universiti Sains Malaysia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IBSXtra02 study
Record Dates: First submitted 2024-10-15; First posted 2024-10-17 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2024-09

CONDITIONS: Irritable Bowel Syndrome (IBS)
Keywords: Irritable Bowel Syndrome (IBS); Synbiotics
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: All study subjects will receive the same study products for 3 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SMT04 Pro (Experimental): 2 sachets daily for 3 months
  Interventions: Dietary Supplement: SMT04 Pro

INTERVENTIONS:
Dietary Supplement: SMT04 Pro — Consists of a blend of food-grade Bifidobacterium as active probiotics

SUMMARY:
Irritable Bowel Syndrome (IBS) is a brain-gut-disorder characterized by a chronic relapsing-remitting nature of symptoms, including abdominal pain and altered bowel habits. Symptoms most likely result from complex interactions between several biological, psychological and social factors.

Probiotic supplements are thought to improve IBS symptoms through manipulation of the gut microbiota. Some studies have suggested that different strains of probiotics may improve abdominal pain and reduce visceral hypersensitivity by modulation of expression of neurotransmitters and receptors involved in the modulation of pain, such as the opioid receptor or the cannabinoid receptor. In addition, probiotics have been shown to reduce intestinal cytokine secretion and improve epithelial barrier function in a mice model of intestinal inflammation.

Bifidobacteria and Streptococci strains had previously demonstrated efficacy in achieving symptom improvement in IBS patients. Thus, there is potential for SMT04, a health supplement, to be an option for IBS patients.

DETAILED DESCRIPTION:
Irritable Bowel Syndrome (IBS) is a common functional bowel disorder characterized by a chronic relapsing-remitting nature of symptoms, including abdominal pain and altered bowel habits. IBS is categorized into four subtypes based on the predominant stool pattern: diarrhoea (IBS-D), constipation (IBS-C), a mix of diarrhoea and constipation (IBS-M) or undefined predominant stool form (IBS-U). The distribution in terms of the predominant stool patterns was IBS-D 37%, IBS-C 27.4%, IBS-M 17.7% and IBS-U 17.7%. Symptoms most likely result from complex interactions between several biological, psychological and social factors and the concept of a brain-gut axis has been evoked.

IBS is a heterogeneous disorder with varying treatments targeted at the predominant symptoms. The optimal approach for any individual can be difficult to determine. Treatment options include both dietary modifications and drug therapies. IBS symptoms are experienced as troublesome for those affected and the condition is associated with increased rates of depression and anxiety, as well as economic challenges, and severe reduction in quality of life (QoL). Neither pharmacological treatment nor diet changes completely eliminate symptoms. Therefore, alternative approaches to improve symptoms and QoL for those affected are needed.

The overall data from gut microbiome research support the approach of adopting novel therapeutic strategies that target the dysbiotic gut for improving gastrointestinal symptoms in IBS. Although probiotic supplements improve IBS symptoms, the precise composition of probiotics that can achieve optimal response remains unclear. SMT04 Pro (GenieBiome (Malaysia) Sdn. Bhd.) is a novel product that is commercially available in Malaysia. It consists of a patented probiotics blend (3 Bifidobacteria, 1 Streptococci, 12.5 billion CFU in 1 sachet). Bifidobacteria and Streptococci strains have been shown to improve in IBS patients. Thus, there is potential for SMT04 Pro, a health supplement, to be an option for IBS patients.

ELIGIBILITY:
Inclusion Criteria:

* The subject must meet all of the inclusion criteria to participate in this study.

  * Male or female,
  * Aged from 18 to 70 years old
  * Meet the criteria of the Rome-III-definition of IBS with diarrhoea or mixed subtypes, or functional diarrhoea: Rome-III-definition: Abdominal pain or abdominal discomfort on minimum of three days per month during the last three months, starting at least six months ago, and a minimum of two of the following criteria:

    * Improvement of symptoms after defecation
    * Start of symptoms in association with a change in stool frequency
    * Start of symptoms in association with a change in stool consistency Subtype of IBS-D which requires more than 25% of your stools to be loose and less than 25% hard and lumpy; Subtype of IBS-M which your stools must be both hard and lumpy, as well as loose in consistency at least 25% of the time. Functional diarrhoea: The experience of loose or watery stools without pain occurring in at least 75% of bowel movements for at least three months over the last six months.
  * Have the latest negative colonoscopy result within five years
  * Literate and can complete questionnaire
  * Written informed consent is obtained

Exclusion Criteria:

* • Known inflammatory bowel disease, lactose intolerance or other malabsorption syndromes, celiac disease, diabetes mellitus, thyroid disfunction, cancer, immunodeficiency, autoimmune diseases, severe hepatic or renal insufficiency, other explainable causes of abdominal pain, diarrhoea or constipation

  * Known operations involving small intestines and large intestines; or history of appendectomy, hysterectomy, and cholecystectomy in last 6 months
  * Known severe mental illnesses; unstable type or dose of psychiatric drugs within the last 3 months that will affect their judgement of study participation
  * Evidence of active infection at the time of inclusion
  * History of use of prebiotics, probiotics, antibiotic therapy or anti-inflammatory drugs within the last 2 weeks
  * Known current pregnancy or breast-feeding female

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-23 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
The improvement of IBS severity using IBS severity scoring system (IBS-SSS) at month 3 after taking SMT04 Pro. | 3 months
  The IBS-SSS score will be used to evaluate the severity of IBS: < 175 for mild IBS, 175-300 for moderate IBS, and > 300 for severe IBS. The higher the score, the worsening of the symptoms.

SECONDARY OUTCOMES:
The change in gastrointestinal symptoms at month 3. | 3 months
  This assessment is to compare the symptom status ranging from XXX to XXX at month 3 compared to baseline. Binary outcome of Yes and No will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Yeong Yeh Lee, Principal Investigator — Universiti Sains Malaysia
Locations (1):
- Universiti Sains Malaysia, Kubang Kerian, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tornkvist NT, Aziz I, Whitehead WE, Sperber AD, Palsson OS, Hreinsson JP, Simren M, Tornblom H. Health care utilization of individuals with Rome IV irritable bowel syndrome in the general population. United European Gastroenterol J. 2021 Dec;9(10):1178-1188. doi: 10.1002/ueg2.12153. Epub 2021 Oct 1. PMID 34599559
- [Background] Mezzasalma V, Manfrini E, Ferri E, Sandionigi A, La Ferla B, Schiano I, Michelotti A, Nobile V, Labra M, Di Gennaro P. A Randomized, Double-Blind, Placebo-Controlled Trial: The Efficacy of Multispecies Probiotic Supplementation in Alleviating Symptoms of Irritable Bowel Syndrome Associated with Constipation. Biomed Res Int. 2016;2016:4740907. doi: 10.1155/2016/4740907. Epub 2016 Aug 9. PMID 27595104
- [Background] Madsen K, Cornish A, Soper P, McKaigney C, Jijon H, Yachimec C, Doyle J, Jewell L, De Simone C. Probiotic bacteria enhance murine and human intestinal epithelial barrier function. Gastroenterology. 2001 Sep;121(3):580-91. doi: 10.1053/gast.2001.27224. PMID 11522742
- [Background] Verdu EF, Bercik P, Verma-Gandhu M, Huang XX, Blennerhassett P, Jackson W, Mao Y, Wang L, Rochat F, Collins SM. Specific probiotic therapy attenuates antibiotic induced visceral hypersensitivity in mice. Gut. 2006 Feb;55(2):182-90. doi: 10.1136/gut.2005.066100. Epub 2005 Aug 16. PMID 16105890
- [Background] Rousseaux C, Thuru X, Gelot A, Barnich N, Neut C, Dubuquoy L, Dubuquoy C, Merour E, Geboes K, Chamaillard M, Ouwehand A, Leyer G, Carcano D, Colombel JF, Ardid D, Desreumaux P. Lactobacillus acidophilus modulates intestinal pain and induces opioid and cannabinoid receptors. Nat Med. 2007 Jan;13(1):35-7. doi: 10.1038/nm1521. Epub 2006 Dec 10. PMID 17159985
- [Background] Jafari E, Vahedi H, Merat S, Momtahen S, Riahi A. Therapeutic effects, tolerability and safety of a multi-strain probiotic in Iranian adults with irritable bowel syndrome and bloating. Arch Iran Med. 2014 Jul;17(7):466-70. PMID 24979556
- [Background] Van den Houte K, Carbone F, Pannemans J, Corsetti M, Fischler B, Piessevaux H, Tack J. Prevalence and impact of self-reported irritable bowel symptoms in the general population. United European Gastroenterol J. 2019 Mar;7(2):307-315. doi: 10.1177/2050640618821804. Epub 2018 Dec 22. PMID 31080615
- [Background] Lea R, Whorwell PJ. New insights into the psychosocial aspects of irritable bowel syndrome. Curr Gastroenterol Rep. 2003 Aug;5(4):343-50. doi: 10.1007/s11894-003-0073-z. PMID 12864966
- [Background] Lovell RM, Ford AC. Global prevalence of and risk factors for irritable bowel syndrome: a meta-analysis. Clin Gastroenterol Hepatol. 2012 Jul;10(7):712-721.e4. doi: 10.1016/j.cgh.2012.02.029. Epub 2012 Mar 15. PMID 22426087
- [Background] El-Salhy M. Irritable bowel syndrome: diagnosis and pathogenesis. World J Gastroenterol. 2012 Oct 7;18(37):5151-63. doi: 10.3748/wjg.v18.i37.5151. PMID 23066308